CLINICAL TRIAL: NCT02589613
Title: Effects of Acute Glucose and Fructose Ingestion on Brain Activity in Obese Volunteers
Brief Title: Glucose and Fructose Stimulated Brain Activity in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: fMRI Obese
Record Dates: First submitted 2015-10-20; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Exploratory Behavior
MeSH Terms: conditions — Exploratory Behavior | interventions — Glucose; Fructose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PLACEBO (Placebo Comparator): Single intragastric instillation of 300ml tap water via nasogastric tube
  Interventions: Dietary Supplement: tap water
- GLUCOSE (Active Comparator): Single intragastric instillation of 75g Glucose in 300ml tap water via nasogastric tube
  Interventions: Dietary Supplement: Glucose
- FRUCTOSE (Active Comparator): Single intragastric instillation of 25g Fructose in 300ml tap water via nasogastric tube
  Interventions: Dietary Supplement: Fructose

INTERVENTIONS:
Dietary Supplement: tap water — 300ml tap water via nasogastric tube
  Arms: PLACEBO
Dietary Supplement: Glucose — 300ml tap water with 75g Glucose via nasogastric tube
  Arms: GLUCOSE
Dietary Supplement: Fructose — 300ml tap water with 25g Fructose via nasogastric tube
  Arms: FRUCTOSE

SUMMARY:
The objective is to investigate neuro-anatomical correlates of the regulation of energy intake by means of functional MRI. Administration of glucose as well as fructose is followed by functional brain MRI, and findings are correlated with serum glucagon-like peptide 1 (GLP-1) levels as an endogenous satiety signal in obese humans.

ELIGIBILITY:
Inclusion Criteria:

* right-handed healthy males, no drugs, non-smoking

Exclusion Criteria:

* drug abuse, smoker, left-handed, claustrophobia

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI) in healthy, obese volunteers while they performed a working memory task: changes in cerebral blood flow | changes from baseline to one hour after treatment

SECONDARY OUTCOMES:
Changes in plasma insulin | changes from baseline to one hour after treatment
Changes in plasma glucose | changes from baseline to one hour after treatment
Changes in plasma GLP-1 | changes from baseline to one hour after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Study Chair — University of Basel